CLINICAL TRIAL: NCT02581176
Title: Apixaban as Treatment of Venous Thrombosis in Patients With Cancer: The CAP Study
Acronym: CAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Anders Dahm, Senior Consultant, Associate Professor, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Neoplasms; Venous Thrombosis
MeSH Terms: conditions — Neoplasms; Venous Thrombosis | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apixaban (Experimental): Apixaban 10 mg two times daily for 1 week, then apixaban 5mg two times daily for 6 months, then apixaban 2.5 mg two times daily for as long as the treating physician finds it necessary.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis

SUMMARY:
This study is a single-arm, phase IV trial, of apixaban as treatment of venous thrombosis in patients with cancer. The current standard treatment of venous thrombosis in cancer patients is subcutaneous injections with low molecular weight heparin. During the last 5 years several new direct acting oral anticoagulants have been tested out as treatment of venous thrombosis. But very few cancer patients were included in the phase III clinical trials of the direct acting oral anticoagulants. Thus, there is a lack of information on how cancer patients with venous thrombosis will respond to treatment with direct acting oral anticoagulants. The current study will investigate the direct acting oral anticoagulant apixaban in cancer patients with venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer, other than basal-cell or squamous-cell carcinoma of the skin, within six months before enrollment. Any treatment for cancer within the previous six months, or recurrent or metastatic cancer.
* Objectively verified venous thrombosis
* Informed consent

Exclusion Criteria:

* Anticoagulant therapy prior to trial entry for > 96 hours
* Severe thrombocytopenia (platelets <50·109/L)
* Severe renal failure - creatinine clearance <30 ml/min
* The patients will be treated with catheter based thrombolysis for deep venous thrombosis or systemic thrombolysis for severe pulmonary embolism
* Pregnancy or breastfeeding.
* Childbearing potential without proper contraceptive measures
* Drug abuse or mental disease that may interfere with treatment and follow-up.
* Severe malabsorption so that oral treatment are expected to have reduced effect
* Mechanical heart valves
* Known allergy to apixaban
* Active bleeding or severe risk of bleeding so that the risk of bleeding is considered a greater danger than the risk of not treating the venous thrombosis
* Clinically significant liver disease (e.g., acute hepatitis, chronic active hepatitis, or cirrhosis)
* Concomitant use of strong cytochrome P-450 3A4 inhibitors (e.g., human immunodeficiency virus protease inhibitors or systemic ketoconazole, voriconazole or posaconazole) or inducers (e.g., rifampicin, carbamazepine, or phenytoin). Fluconazol is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Recurrent objectively confirmed venous thrombosis or death related to venous thrombosis | 6 months after inclusion
Major or clinically relevant non-major bleeding | 6 months after inclusion

SECONDARY OUTCOMES:
All cause mortality | 6 months after inclusion
All cause mortality | 24 months after inclusion
Recurrent objectively confirmed venous thrombosis or death related to venous thrombosis | 24 months after inclusion
Major or clinically relevant non-major bleeding | 24 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Anders EA Dahm, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (9):
- Norway (9):
  - Haukeland University Hospital, Bergen
  - Vestre Viken- Drammen Hospital, Drammen
  - Vestre Viken - Bærum sykehus, Gjettum
  - Department of Hematology, Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Østfold Hospital Kalnes, Sarpsborg
  - Stavanger University Hospital, Stavanger
  - St. Olavs Hospital, Trondheim
  - Volda Hospital, Volda

REFERENCES:
- [Derived] Larsen TL, Svalastoga M, Brekke J, Enden T, Froen H, Garresori H, Jacobsen EM, Paulsen PQ, Porojnicu AC, Ree AH, Torfoss D, Velle EO, Wik HS, Ghanima W, Sandset PM, Dahm AEA. Arterial events in cancer patients treated with apixaban for venous thrombosis. Thromb Res. 2023 Aug;228:128-133. doi: 10.1016/j.thromres.2023.05.017. Epub 2023 May 25. PMID 37327527
- [Derived] Hannevik TL, Brekke J, Enden T, Froen H, Garresori H, Jacobsen EM, Paulsen PQ, Porojnicu AC, Ree AH, Torfoss D, Velle EO, Wik HS, Ghanima W, Sandset PM, Dahm AEA. Thrombosis and bleedings in a cohort of cancer patients treated with apixaban for venous thromboembolism. Thromb Res. 2020 Dec;196:238-244. doi: 10.1016/j.thromres.2020.08.042. Epub 2020 Aug 28. PMID 32919178